CLINICAL TRIAL: NCT04570852
Title: Acute Pancreatitis Targets (APT) Study
Acronym: APT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, John Gasdal Karstensen, Associate professor, MD, PhD, Copenhagen University Hospital, Hvidovre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APT
Record Dates: First submitted 2020-09-22; First posted 2020-09-30 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Pancreatitis, Acute
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intensive monitoring of patients (Experimental): State of the art biochemical assessment of patients with acute pancreatitis including multi-OMICS focusing on transcriptomics and proteomics.
  Interventions: Other: LiDCO

INTERVENTIONS:
Other: LiDCO — We plan to elucidate the pathophysiology and molecular subtypes of acute pancreatitis in order to develop specific biomarkers and identify new drug targets. The evaluation will include an analysis of the impact of obesity and the metabolic profile during the disease course of acute pancreatitis.
  Supportive treatments will be registered including an assessment of the fluid balance based on the fluid intake and loss and weight. Bioimpedance will be assessed at admission/day1, day 2, day 3,
  Other Names: Bioimpedance; Ommics; Rutine blood samples; TEQ

SUMMARY:
The severity of acute pancreatitis varies considerably from minor symptoms to multi-organ failure. The pathophysiological mechanisms associated with these individual differences in severity are largely unknown. Acute pancreatitis is therefore classified based on clinical characteristics and routine blood samples. Information about pathophysiology and molecular subtypes of acute pancreatitis is needed to develop specific biomarkers and identify new drug targets. The investigators therefore plan to undertake an explorative study, which includes state-of-the-art biochemical assessment of patients with acute pancreatitis including multi-OMICS focusing on transcriptomics and proteomics.

DETAILED DESCRIPTION:
Introduction Acute pancreatitis is a sudden inflammation of the pancreas with clinical manifestations ranging from a mild self-limiting disease to a severe form with necrosis of the pancreas and multi-organ dysfunction. Population-based cohort studies report a global incidence of 23 to 49 cases per 100,000 per year. In Denmark, more than 4,000 patients are admitted with acute pancreatitis each year. Gallstones and alcohol account for approximately 80% of all cases. Although the clinical characteristics and induction mechanism differ in the two groups, no differences in the inflammatory profile have been identified.

Acute pancreatitis is characterised by an early phase 7-10 days after the onset and a late phase after more than 10-14 days. The early phase is dominated by the host response to the local pancreatic injury leading to systemic inflammation. The late phase is characterized by infected pancreatic or peri-pancreatic necrosis, systemic signs of infection, and possible local complications including splanchnic vein thrombosis. Multi-organ dysfunction may occur in the early as well as the late phase. Although supportive treatment and minimally invasive techniques have improved the overall prognosis, the mortality among patients with severe pancreatitis remains about 10 to 15%. Once persistent multi-organ dysfunction develops, mortality is as high as 30 to 40%.

Following an episode of acute pancreatitis patients are in risk of developing comorbidities. Fifteen percent of the patients will develop diabetes within a year and 10 % will develop chronic pancreatitis after a first episode of acute pancreatitis.

At present time, there are no specific treaments to prevent attacks of acute pancreatitis, nor there are any disease modifying measures. Patients are mainly treated with supportive care which includes close monitoring of organ functions, pain management, fluid resuscitation and nutrition.

Several prognostics scores have been developed to identify patients at risk of developing severe acute pancreatitis. The scores are used in patient triage. Most scores include age and an assessment of the respiratory, circulatory and renal function. Blood glucose, platelets, albumin and calcium are used as markers of third space fluid losses, inflammation, lipolysis/fat necrosis and impaired pancreatic endocrine function. Other clinical variables include obesity, body mass index (BMI) and abdominal fat.

Genetic polymorphisms in the tumour necrosis factor (TNF)-alfa and the Monocyte chemoattractant protein (MCP)-1 genes are associated with an increased risk of acute pancreatitis, but none are currently used in clinical practice.

Pancreatic enzymes Activation of the pancreatic enzymes: amylase, lipases (including pancreatic lipase, phospholipase and sterol esterase) and proteases (including trypsin, chymotrypsin, carboxypeptidase and elastases) play a key role in the development of acute pancreatitis. Elevated amylase and lipase are used in the diagnosis, but cannot predict disease severity.

Trypsin and elastase levels are elevated for a longer time than amylase and lipase along with their potential catalysing effects on proteins.

Locally, activated enzymes are responsible for the development of pancreatic and peripancreatic necrosis, but little is known about the effect of the circulating enzymes. Theoretically, the enzymes can catalyse degradation of carbohydrates, lipids and protein throughout the body causing systemic metabolic alterations and contribute to disease severity and progression.

Endocrine function Acute pancreatitis is associated with extensive metabolic changes, which occur from the early stage. Elevated plasma glucose is used as a predictor of the disease severity. Possibly hyperglycaemia worsens the outcome, but also could be a marker of pancreatic damage and the metabolic stress related to critical illness. Hyperglycaemia on admission was associated with the development of pancreatic necrosis and pseudocysts and longer hospital stay The findings regarding hyperglycaemia organ dysfunction are equivocal.

Patients with acute pancreatitis have increased degradation of pro, but also increased proinsulin and insulin levels as well as glucagon and glucagon related peptides during the first days after hospital admission. The levels are fluctuating and may reflect a combination of a transient reduction in secretion from beta-cells and changes in the breakdown by activated proteases from the pancreas.

Increased levels of cortisol during the acute inflammatory acute phase are also likely to be involved in the metabolic changes. The studies investigating endocrine function during acute pancreatitis are limited and only include few patients.

The complex interactions between inflammatory pathways, gut hormones, obesity and endocrine function is impaired even after the initial stage of the inflammatory disease.

Obesity, lipolysis and acute pancreatitis In patients with acute pancreatitis, obesity is associated with the risk of both local and systemic complication. Theoretically, obesity-associated low-grade inflammatory predisposes to the development of a systemic inflammatory response. Serum concentrations of interleukins and c-reactive protein (CRP) were increased in patients with obesity, and adiponectin levels are associated with the severity of acute pancreatitis. Furthermore, abdominal adiposity increases the risk of acute pancreatitis and is correlated with the severity, local complications and death. The association may reflect lipolysis in the visceral adipose tissue and the concentration of fatty acids is increased in pancreatic necrotic collections. Intraperitoneal administration of unsaturated fatty acids to rats in a model of acute pancreatitis, increased cytokine levels was associated with an increased risk of multi-organ dysfunction, pancreatic necrosis and mortality. These changes were prevented by the administration of the lipase inhibitor orlistat.

Proteomics and acute pancreatitis Previous studies have assessed the identity and amount of proteins as well as proteolysis and post-translational modifications of proteins in acute pancreatitis. Animal models have found an increase in certain proteins related to stress and inflammation. The increase can occur through an increased synthesis as well as migration or decreased degradation. Similar changes are likely to occur in humans. Transcriptomic profiling has not been performed in acute pancreatitis. However, the method has provided invaluable information about inflammatory changes, potential diagnostic markers and cellular changes in several different diseases such as diabetes, non-alcoholic fatty liver disease and pancreatic cancer.

Objective The investigators plan to elucidate the pathophysiology and molecular subtypes of acute pancreatitis in order to develop specific biomarkers and identify new drug targets. The evaluation will include an analysis of the impact of obesity and the metabolic profile during the disease course of acute pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age >18 years) with acute pancreatitis according to the revised Atlanta criteria;12
* Informed consent;
* Known time of debut of symptoms.

Exclusion Criteria:

* Chronic pancreatitis;
* Pregnancy;
* Known malignant disease;
* More than 72 hours from debut of symptoms to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with severe pancreatitis | 90 days
  Development og severe pancreatitis according to standard definitions

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenheden, Hvidovre Hospital, Hvidovre, Capital, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Background] Xiao AY, Tan ML, Wu LM, Asrani VM, Windsor JA, Yadav D, Petrov MS. Global incidence and mortality of pancreatic diseases: a systematic review, meta-analysis, and meta-regression of population-based cohort studies. Lancet Gastroenterol Hepatol. 2016 Sep;1(1):45-55. doi: 10.1016/S2468-1253(16)30004-8. Epub 2016 Jun 28. PMID 28404111
- [Background] Landspatientregisteret. Datatræk på "Akut pankreatitis". Tilgået 6 juni 2019. Tilgængelig via: esundhed.dk.
- [Background] Novovic S, Andersen AM, Ersboll AK, Nielsen OH, Jorgensen LN, Hansen MB. Proinflammatory cytokines in alcohol or gallstone induced acute pancreatitis. A prospective study. JOP. 2009 May 18;10(3):256-62. PMID 19454816
- [Background] Mofidi R, Duff MD, Wigmore SJ, Madhavan KK, Garden OJ, Parks RW. Association between early systemic inflammatory response, severity of multiorgan dysfunction and death in acute pancreatitis. Br J Surg. 2006 Jun;93(6):738-44. doi: 10.1002/bjs.5290. PMID 16671062
- [Background] van Santvoort HC, Bakker OJ, Bollen TL, Besselink MG, Ahmed Ali U, Schrijver AM, Boermeester MA, van Goor H, Dejong CH, van Eijck CH, van Ramshorst B, Schaapherder AF, van der Harst E, Hofker S, Nieuwenhuijs VB, Brink MA, Kruyt PM, Manusama ER, van der Schelling GP, Karsten T, Hesselink EJ, van Laarhoven CJ, Rosman C, Bosscha K, de Wit RJ, Houdijk AP, Cuesta MA, Wahab PJ, Gooszen HG; Dutch Pancreatitis Study Group. A conservative and minimally invasive approach to necrotizing pancreatitis improves outcome. Gastroenterology. 2011 Oct;141(4):1254-63. doi: 10.1053/j.gastro.2011.06.073. Epub 2011 Jul 8. PMID 21741922
- [Background] Johnson CD, Abu-Hilal M. Persistent organ failure during the first week as a marker of fatal outcome in acute pancreatitis. Gut. 2004 Sep;53(9):1340-4. doi: 10.1136/gut.2004.039883. PMID 15306596